CLINICAL TRIAL: NCT02512133
Title: MIGS VS SLT in Glaucoma Patients: Prospective Study
Brief Title: MIGS VS SLT Comparison in Glaucoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: University of Siena (Other)
Responsible Party: Principal Investigator, Antonio Fea, Aggregate Professor, University of Turin, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-07-19; First posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Glaucoma
Keywords: MIGS; SLT
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIGS Hydrus Ivantis (Experimental): opening the anterior chamber (2mm.) injecting visco-material, injecting the Hydrus stent in the Schlemm's canal under gonioscopic control
  Interventions: Device: MIGS Hydrus Ivantis
- SLT (Experimental): Laser Solutis SLT laser (Quantel Medical, Clermont-Ferrand, France): this frequency-doubled, Q-switched Nd:YAG laser emits light at a wavelength of 532 nm, with a pulse duration of 4 ns, a spot size of 400 µm and pulse energy ranging from 0.2 to 2 mJ
  Interventions: Procedure: 360 degrees SLT

INTERVENTIONS:
Device: MIGS Hydrus Ivantis — implant of the micro stent in the nasal Schlemm's canal
  Arms: MIGS Hydrus Ivantis
Procedure: 360 degrees SLT — Laser Solutis SLT laser (Quantel Medical, Clermont-Ferrand, France): this frequency-doubled, Q-switched Nd:YAG laser emits light at a wavelength of 532 nm, with a pulse duration of 4 ns, a spot size of 400 µm and pulse energy ranging from 0.2 to 2 mJ
  Arms: SLT

SUMMARY:
To compare the intraocular pressure (IOP) and number of glaucoma medications lowering of microinvasive glaucoma surgery (MIGS) with the implantation of the trabecular device Hydrus (Ivantis) as a solo procedure and 360° selective laser trabeculoplasty (SLT) to treat primary open angle glaucoma (POAG).

DETAILED DESCRIPTION:
Eligible study patients diagnosed with POAG and not sufficiently controlled by, intolerant of, or non-compliant with their current IOP-lowering regimen. Patients with IOP>21 mm Hg upon at least two consecutive measurements. Study subjects with typical glaucomatous visual field (VF) loss on Octopus or Humphrey automated perimetry (Carl Zeiss Meditec, Dublin, CA) and glaucomatous alterations to the optic nerve head. Visual field classified as glaucomatous according to the European Glaucoma Society guidelines.

Exclusion criteria : eye surgery in the previous 6 months, any previous surgery for glaucoma, evidence of glaucoma of a type other than POAG, and medication with systemic or topical steroids.

ELIGIBILITY:
Inclusion Criteria:

* primary open angle glaucoma diagnosis, intolerant or unresponsive to therapy or not controlled with therapy

Exclusion Criteria:

* eye surgery in the previous 6 months, any previous surgery for glaucoma, evidence of glaucoma of a type other than POAG, and medication with systemic or topical steroids

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2014-04 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
change in the intraocular pressure compared to baseline | up to 12 months
  measurement with GAT in mm Hg

SECONDARY OUTCOMES:
change in the number of glaucoma medications compared to baseline | up to 12 months
  accountability of IOP lowering medications used by the patient

OTHER OUTCOMES:
change of visual acuity compared to baseline | 6 months and 1 year post-intervention
  ETDRS visual acuity scale
change of visual field compared to baseline | 1 year post-intervention
  MD and PSD

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fea, MD, Principal Investigator — Clinica Oculistica
Locations (1):
- Ophthalmology Institute, University of Turin, Turin, Italy

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114